CLINICAL TRIAL: NCT07307274
Title: A Phase 1 Randomised, Double-blind, Placebo-controlled Single Ascending and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SYNT-101 in Healthy Adults and Healthy Adults Who Are Overweight or Have Obesity
Brief Title: A Study of SYNT-101 to Test Safety, Tolerability and Pharmacodynamics of SYNT-101 in Healthy and Overweight Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Syntis Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SYNT101-001
Record Dates: First submitted 2025-11-27; First posted 2025-12-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Overweight and Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Drug SYNT101 (Active Comparator)
  Interventions: Drug: SYNT101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYNT101 — Tablet
  Arms: Active Drug SYNT101
Drug: Placebo — Placebo tablet to match SYNT101 in appearance.
  Arms: Placebo

SUMMARY:
A Phase 1, single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacodynamics of single and multiple dose regimens of SYNT-101 in healthy and overweight adults.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
* Adult males and females, 18 to 55 years of age (inclusive) at screening.
* Medically healthy (in the opinion of the PI or delegate), as determined by pre-study medical history, and without clinically significant (CS) abnormalities.
* Have suitable venous access for blood sampling.
* Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

* Known hypersensitivity to the study drug or any of the study drug ingredients.
* History of anaphylaxis or other significant allergy which, in the opinion of the PI (or delegate), would interfere with the volunteer's ability to participate in the study.
* History or presence of CS cardiovascular, pulmonary, hepatic, renal, haematological, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder, including any acute illness, within the past 3 months determined by the PI (or delegate) to be clinically relevant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation | From enrolment up to 7 days post dosing in the SAD and up to 36 days post dosing in the MAD.
  The Number of participants with Adverse Events, with abnormal Vital Signs, abnormal Physical Examination findings, abnormal Laboratory Tests results, abnormal 12-lead Electrocardiogram (ECG) readings.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) after single SYNT101 dose | At Pre-dose, 1 hr , 3 hr, 4 hr, 8 hr, 12 hr, 24 hours post-dose.
  Evaluate the pharmacokinetics (Area Under the Plasma Concentration Curve) of SYNT101 after a single dose via measuring concentration levels in the blood.
Area under the plasma concentration versus time curve (AUC) after multiple SYNT101 doses. | At Pre-Dose, 1 hr , 3 hr, 4 hr, 8 hr, 12 hr, 24 hours post-dose.
  Evaluate the pharmacokinetics (Area Under the Plasma Concentration Curve) of SYNT101 after multiple doses via measuring concentration levels in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Veritus Research, Bayswater, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No